CLINICAL TRIAL: NCT04364191
Title: Multicomponent Behavioral Sleep Intervention for Insomnia in Older Adults With Mild Cognitive Impairment
Acronym: MBSI-I
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 832826; K23NR018487 (NIH)
Record Dates: First submitted 2020-04-15; First posted 2020-04-28 (Actual); Results first posted 2024-05-29 (Actual); Last update posted 2024-05-29 (Actual); Status verified 2024-05

CONDITIONS: Mild Cognitive Impairment; Insomnia
MeSH Terms: conditions — Cognitive Dysfunction; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Arm (Experimental): Meaningful activity protocol during the day and Assisted Relaxation Therapy (ART) at night; includes 1) Sleep Hygiene Education; 2) Meaningful Activity Modules a) Physical Activity b) Cognitive Activity and c) Social engagement; 3) ART, a breath-based relaxation intervention that is coupled with a physical anchoring task. Participants will complete a daily sleep diary, use the activity modules daily as pre-determined times personalized to the participant, use the ART software when they get in bed to help with insomnia symptoms, and wear an actiwatch for a four-week period. Participants will have weekly to biweekly phone consultation with the research nurse.
  Interventions: Behavioral: Multicomponent Behavioral Sleep Intervention for Insomnia
- Control Arm (Active Comparator): Study participants in the control group will also receive a tablet and watch, but the meaningful activity modules and ART software will not be accessible to them. The sleep hygiene educational material represents an active control intervention and is recommended as part of the initial treatment of insomnia based on an NIH guide for sleep education. This approach provides staff and technology interaction/attention that is comparable to the intervention arm, and thereby promotes adherence; it has been used as a placebo comparator for many insomnia treatment studies and has low attrition rates. Control subjects will also be asked to complete electronic sleep diaries and wear the actiwatch on the non-dominant wrist to monitor sleep/wake patterns. For both arms, participants will be asked to complete baseline assessments, 4-week (post-intervention) and 12-week (follow-up).
  Interventions: Behavioral: Active Control

INTERVENTIONS:
Behavioral: Multicomponent Behavioral Sleep Intervention for Insomnia — The MBSI-I will include a meaningful activity protocol during the day and ART therapy at night.
  Arms: Intervention Arm
Behavioral: Active Control — The sleep hygiene educational material represents an active control intervention and is recommended as part of the initial treatment of insomnia based on an NIH guide for sleep education.
  Arms: Control Arm

SUMMARY:
Insomnia symptoms in older adults with mild cognitive impairment represent a significant public health burden in terms of impaired quality of life, risks from untreated insomnia, and risks from pharmaceutical insomnia treatment. To address the limitations in the most effective non-pharmacological treatments for insomnia in older adults with mild cognitive impairment, a randomized pilot study will be conducted to test a brief (4 week), tablet-based, personalized, multicomponent behavioral sleep intervention for insomnia, compared to a sleep education control, in this at-risk group. The findings of the proposed project will inform future, larger scale clinical trials and may provide a novel and innovative way for older adults with mild cognitive impairment to achieve better sleep and health-related quality of life outcomes.

ELIGIBILITY:
Inclusion Criteria:

* 1) age 55 and older
* 2) mild cognitive impairment (MCI) The Telephone Interview for Cognitive Status 13-item modified (TICS-M) version will be used to screen participants for eligibility in the study. We will include participants with TICS-M scores of 28-36, based off ranges and optimal cutpoints determined in various studies.
* 3) have insomnia symptoms a)answer yes to "Do you have trouble falling asleep, staying asleep, awakening too early, or have unrefreshing sleep" and b) have subjective sleep diary evidence of insomnia, with an average sleep onset latency >30 min or wakefulness after sleep onset of >60 min during the one week pre-treatment assessment
* 4) live in the community
* 5) speak English as primary language

Exclusion Criteria:

* 1) Presence of moderate to severe cognitive impairment defined as TICS score <28
* 2) Visual or manual dexterity impairment that prevents them from pressing yes/no buttons, or selecting a number at 24 point font
* 3) Current sedative-hypnotic or other sleep aid use on a regular or as needed schedule within the prior three months
* 4) Presence of an acute medical or psychiatric condition which, in the judgement of the research team, would interfere with the subject's ability to realistically follow the study protocol

Min Age: 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2021-05-13 (Actual); Primary Completion 2022-08-30 (Actual); Study Completion 2022-08-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Screened 180 participants
Period: Overall Study
Arm/Group | Intervention Arm | Control Arm
Started | 13 | 14
Completed | 12 | 12
Not Completed | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention Arm | Control Arm | Total
Number analyzed (Participants) | 13 | 14 | 27
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.93 (7.13) | 65.31 (5.75) | 65.63 (6.39)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 12 | 22
  Male | 3 | 2 | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 13 | 13 | 26
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 7 | 12
  White | 8 | 6 | 14
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0
subjective sleep latency [Mean (Standard Deviation); unit: minutes] — The time that it takes someone to fall asleep, from the first intention of going to sleep, in minutes. This variable is collected via sleep diary and averaged over a one week period.
  minutes | 41.42 (33.10) | 46.57 (27.73) | 44.09 (29.95)
subjective sleep efficiency [Mean (Standard Deviation); unit: percentage] — The percentage of time spent in bed that a person actually is asleep (time asleep/time in bed). This variable is collected via sleep diary and averaged over a one week period.
  percentage | 70 (12) | 65 (11) | 67.90 (11.94)
subjective total sleep time [Mean (Standard Deviation); unit: minutes] — The amount of time a person is asleep at night. This variable is collected via sleep diary and averaged over a one week period.
  minutes | 346.27 (85.42) | 336.00 (64.54) | 341.14 (74.36)
subjective wake after sleep onset [Mean (Standard Deviation); unit: minutes] | 44.85 (28.38) | 46.30 (40.56) | 45.63 (34.79)
36-Item Short Form Survey (SF-36) [Mean (Standard Deviation); unit: units on a scale] — RAND Medical Outcomes Study Short Form-36 (SF-36) is a multidomain scale that measures physical and mental components of HRQOL with eight subscales. The 8 subscales include physical functioning, bodily pain, role limitations due to physical health problems, role limitations due to personal or emotional problems, general mental health, social functioning, energy/fatigue, and general health and range from 0 to 100 (lower scores indicate worse HRQOL). For this primary analysis, we are using the general health scale.
  units on a scale | 59.23 (34.02) | 58.93 (21.41) | 59.07 (27.63)
Insomnia Severity Index [Mean (Standard Deviation); unit: scores on a scale] — The ISI is a validated self-report measure of insomnia. Participants answer 7 questions; scores are summed. Scores range from 0-28; higher scores indicate worse sleep (I.e., more insomnia).
  scores on a scale | 13.23 (4.17) | 14.5 (4.80) | 13.89 (4.47)
Pittsburgh Sleep Quality Index [Mean (Standard Deviation); unit: score on a scale] — This is a validated measure of self-reported sleep quality. The measure consists of 19 individual items, creating 7 components that produce one global score. Higher scores indicate worse sleep quality.
  score on a scale | 9.85 (2.61) | 10.86 (2.63) | 10.37 (2.62)
Number of Participants who Completed the Dried Blood Spot Sample for Inflammatory Biomarker Analysis [Count of Participants; unit: Participants] — this measure was a count of participants who completed the dried blood spot collections to be used for inflammatory biomarker analysis and is being used as a feasibility measure.
  Participants | 11 | 9 | 20

OUTCOME MEASURES:

1. Primary Outcome: Sleep Latency
Description: time it takes a person to fall asleep, starting from first intention to sleep, measured by sleep diary
Time Frame: immediately post-intervention (4-5weeks after the start of the intervention)
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Intervention Arm | Control Arm
Number analyzed (Participants) | 12 | 13
minutes | 28.51 (31.18) | 47.06 (34.61)

2. Primary Outcome: Sleep Latency
Description: time it takes a person to fall asleep, starting from first intention to sleep; measured by sleep diary
Time Frame: 3 months post intervention
Population: Lost one participant in intervention to follow-up; lost two participants in control arm to follow up and one had missing sleep diary data at follow up
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Intervention Arm | Control Arm
Number analyzed (Participants) | 12 | 11
minutes | 25.39 (27.02) | 35.92 (32.44)

3. Primary Outcome: Health Related Quality of Life (HRQOL)
Description: RAND Medical Outcomes Study Short Form-36 (SF-36) is a multidomain scale that measures physical and mental components of HRQOL with eight subscales. The 8 subscales include physical functioning, bodily pain, role limitations due to physical health problems, role limitations due to personal or emotional problems, general mental health, social functioning, energy/fatigue, and general health. All sub scales range from 0 to 100 (lower scores indicate worse HRQOL). For this primary analysis, we are using the general health sub scale, ranging from 0 to 100, where lower scores indicate worse HRQOL.
Time Frame: immediately post-intervention (4-5weeks after the start of the intervention)
Population: lost one intervention participant and one control participant to immediate follow up
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention Arm | Control Arm
Number analyzed (Participants) | 12 | 13
score on a scale | 60.83 (31.10) | 58.08 (20.97)

4. Primary Outcome: Health Related Quality of Life (HRQOL)
Description: as for outcome 3
Time Frame: 3 months post intervention
Population: Lost one participant to immediate follow-up in intervention group and one to immediate follow-up in control and one at 3 mo follow up in control group.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention Arm | Control Arm
Number analyzed (Participants) | 12 | 12
score on a scale | 55.83 (29.99) | 54.58 (22.71)

5. Secondary Outcome: Wake After Sleep Onset (WASO)
Description: time (in minutes) a person spends awake during the night, starting from the time the person falls asleep; derived from actigraphy monitoring; more WASO indicates worse sleep
Time Frame: immediately post intervention (4-5weeks after the start of the intervention)
Population: lost one intervention participant and one control participant to immediate follow up
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Intervention Arm | Control Arm
Number analyzed (Participants) | 12 | 13
minutes | 29.57 (33.70) | 37.25 (32.49)

6. Secondary Outcome: Wake After Sleep Onset (WASO)
Description: as for outcome 5
Time Frame: 3 months post intervention
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Intervention Arm | Control Arm
Number analyzed (Participants) | 12 | 12
minutes | 29.30 (33.06) | 35.21 (43.57)

7. Secondary Outcome: Total Sleep Time (TST)
Description: Actual time (in minutes) a person is asleep during the nighttime sleep period; derived from actigraphy monitoring; normal sleep ranges from 420-480 minutes
Time Frame: immediately post intervention
Population: lost one intervention participant and one control participant to immediate follow up
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Intervention Arm | Control Arm
Number analyzed (Participants) | 12 | 13
minutes | 368.78 (90.03) | 361.43 (70.86)

8. Secondary Outcome: Total Sleep Time (TST)
Description: as for outcome 7
Time Frame: 3 months post intervention
Population: Lost one participant to immediate follow-up in intervention group and one to immediate follow-up in control and one at 3 mo follow up in control
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Intervention Arm | Control Arm
Number analyzed (Participants) | 12 | 12
minutes | 381.38 (70.46) | 340.38 (90.11)

9. Secondary Outcome: Sleep Efficiency (SE)
Description: Percent of time spent in bed that a person is asleep; calculated from actigraphy (time asleep/ time in bed)x 100%; lower SE indicates worse sleep
Time Frame: immediately post intervention
Population: lost one intervention participant and one control participant to immediate follow up
Measure: Mean (Standard Deviation); unit: percentage of time asleep
Arm/Group | Intervention Arm | Control Arm
Number analyzed (Participants) | 12 | 13
percentage of time asleep | 77 (12) | 68 (14)

10. Secondary Outcome: Sleep Efficiency (SE)
Description: as for outcome 9
Time Frame: 3 months post intervention
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: percentage of time spent asleep
Arm/Group | Intervention Arm | Control Arm
Number analyzed (Participants) | 12 | 12
percentage of time spent asleep | 77 (13) | 66 (17)

11. Secondary Outcome: Self- Reported Insomnia Symptoms
Description: measured with the Insomnia Severity Index; score ranges from 0-28, with higher scores indicating more insomnia symptoms (thus worse outcomes)
Time Frame: immediately post intervention
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention Arm | Control Arm
Number analyzed (Participants) | 12 | 13
score on a scale | 12 (10.67) | 12.5 (4.75)

12. Secondary Outcome: Self- Reported Insomnia Symptoms
Description: as for outcome 11
Time Frame: 3 months post intervention
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention Arm | Control Arm
Number analyzed (Participants) | 12 | 12
score on a scale | 9.42 (4.21) | 11.83 (4.86)

13. Secondary Outcome: Self-reported Sleep Quality
Description: measured with Pittsburgh Sleep Quality Index; score ranges from 0-21 with higher scores indicating poor sleep quality (worse outcomes)
Time Frame: immediately post intervention
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention Arm | Control Arm
Number analyzed (Participants) | 12 | 13
score on a scale | 8.83 (2.68) | 10.29 (2.76)

14. Secondary Outcome: Self-reported Sleep Quality
Description: as for outcome 13
Time Frame: 3 months post intervention
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention Arm | Control Arm
Number analyzed (Participants) | 12 | 12
score on a scale | 8.5 (2.68) | 10.17 (1.75)

15. Other Pre Specified Outcome: Number of Participants Who Completed the Dried Blood Spot Sample for Inflammatory Biomarker Analysis
Description: Systemic inflammatory markers will be assayed using dried blood spots (DBS). DBS provides an easy to obtain, transport, and analyze blood source. Our Translational Core Laboratory utilizes a matrix independent platform (Mesoscale Discovery, Rockville MD), to support the assay of DBS for systemic inflammatory markers. Participants who have trouble with the finger prick will be provided with verbal assistance at sample pick-up while the researcher maintains physical distance. The outcome measure used for this study will be number of participants who complete the dried blood spot sample, as a measure of feasibility.
Time Frame: Immediately post intervention
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Arm | Control Arm
Number analyzed (Participants) | 12 | 13
Participants | 10 | 4

16. Other Pre Specified Outcome: Number of Participants Who Completed the Dried Blood Spot Sample for Inflammatory Biomarker Analysis
Description: Systemic inflammatory markers will be assayed using dried blood spots (DBS). DBS provides an easy to obtain, transport, and analyze blood source. Our Translational Core Laboratory utilizes a matrix independent platform (Mesoscale Discovery, Rockville MD), to support the assay of DBS for systemic inflammatory markers. Participants who have trouble with the finger prick will be provided with verbal assistance at sample pick-up while the researcher maintains physical distance.
Time Frame: 3 months post intervention
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Arm | Control Arm
Number analyzed (Participants) | 12 | 13
Participants | 8 | 6

ADVERSE EVENTS:
Time Frame: Adverse event data were collected at each touchpoint with participant- Weekly during the intervention, visit 2 (5 weeks after baseline), Visit 3 (17 weeks after baseline)
Description: No difference
Arm/Group | Intervention Arm | Control Arm
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/14
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/14
Other Adverse Events (participants affected / at risk) | 0/13 | 0/14

LIMITATIONS AND CAVEATS:
Dried blood spot analysis was changed into a feasibility measure, given the low responses.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-03-15): https://cdn.clinicaltrials.gov/large-docs/91/NCT04364191/Prot_SAP_004.pdf
  • Informed Consent Form (2021-03-30): https://cdn.clinicaltrials.gov/large-docs/91/NCT04364191/ICF_003.pdf